CLINICAL TRIAL: NCT01936402
Title: Novel Instruction to Perform Chest Compression Approximately 6-7cm for Healthcare Provider Improves Chest Compression Depth During Cardiopulmonary Resuscitation in Hospital.
Brief Title: Instruction to Compress Chest Approximately 6-7cm for Healthcare Provider in Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaehoon Oh (Other)
Responsible Party: Sponsor-Investigator, Jaehoon Oh, Emergency department, Hanyang University
Organization: Hanyang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CCD5565
Record Dates: First submitted 2013-08-29; First posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Cardiac Arrest
Keywords: Cardiopulmonary Resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-6cm Chest compression depth (Experimental): Control group is trained for 5-6cm Chest compression depth during education.
  Depth 5-6cm, Rate 100-120/min, Full chest recoil
  Interventions: Behavioral: Education of chest compression depth
- 6-7cm chest compression depth (Experimental): Experimental group is trained for 6-7cm Chest compression depth during education.
  Depth 6-7cm, Rate 100-120/min, Full chest recoil
  Interventions: Behavioral: Education of chest compression depth

INTERVENTIONS:
Behavioral: Education of chest compression depth — An American Heart Association Basic Life Support faculty educated each participant in Experimental group a standard 30-min lecture and hands- on practice for chest compression without ventilation using manikin on the floor according to 5-6cm or 6-7cm chest compression depth

SUMMARY:
Unlikely the other element for high quality chest compression during Cardiopulmonary resuscitation(i.e. compression rate, chest recoil, hand position), chest compression depth (CCD) is influenced by surface on which the patient is placed, especially in hospital. For solving this problem, to place the patient on rigid surface, use a backboard that might decrease the mattress compression, receive a feedback that reflects the mattress compression depth (MCD) using dual accelerometer or magnetic sensor have been proposed. As the other solution, we hypothesized that training of 6-7cm CCD for healthcare providers improve accurate CCD during cardiopulmonary resuscitation when manikin is placed on mattress in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Medical students, Healthy

Exclusion Criteria:

* Heart, wrist, and low back disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change of Chest compression depth at 4 weeks | 1 hour and 4weeks later after education

SECONDARY OUTCOMES:
Change of Chest compression rate at 4 weeks | 1 hour and 4weeks later after education

OTHER OUTCOMES:
Change of number of Chest decompression at 4 weeks | 1 hour and 4weeks later after education